CLINICAL TRIAL: NCT06088160
Title: Changes in Postural Stability and Balance Confidence in People After Elective Unilateral Total Hip Arthroplasty for Osteoarthritis: A Prospective Cohort Study
Brief Title: Changes in Postural Stability Following THA for OA
Acronym: CPS
Status: Recruiting | Type: Observational
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 123634
Record Dates: First submitted 2023-09-28; First posted 2023-10-18 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis, Hip
Keywords: Postural stability; Total hip arthroplasty; Balance confidence; Osteoarthritis; Fall
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Direct Anterior: This group will consist of people undergoing elective unilateral THA for OA using the Direct Anterior surgical approach
  Interventions: Procedure: Total Hip Arthroplasty
- Direct Lateral: This group will consist of people undergoing elective unilateral THA for OA using the Direct Lateral surgical approach
  Interventions: Procedure: Total Hip Arthroplasty

INTERVENTIONS:
Procedure: Total Hip Arthroplasty — Total hip arthroplasty is a common surgical procedure performed in people with advanced hip osteoarthritis
  Other Names: Total hip replacement

SUMMARY:
Total hip arthroplasty (THA) is a common surgery that eases pain, restores functional movement, and improves the overall quality of life in people with severe hip osteoarthritis (OA). Unfortunately, problems with postural stability, commonly known as balance, are still noticed in people even years after the surgery. These postural stability problems typically result in falls. The aim of the proposed study is to investigate how THA surgery affects a person's overall quality of life, both physically and psychologically, in terms of postural stability and balance confidence (self-efficacy) within the first three months after THA for osteoarthritis. This prospective cohort study will focus on people over 60 years old.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the changes in postural stability and balance confidence during the initial three months after elective unilateral total hip arthroplasty for osteoarthritis. Specifically, the investigators aim to:

1. To evaluate change in postural stability between the DA and DL surgical approaches during the first three months after elective unilateral THA for OA, using both a clinical measure and an instrumented measure.
2. To evaluate change in balance confidence between the DA and DL surgical approaches during the first three months after elective unilateral THA for OA.

   Secondary objective
3. To compare the DA and DL approaches for activity levels, function, quality of life and pain during the first three months after elective unilateral THA for OA.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 60 years of age, scheduled to receive an elective unilateral THA (DA or DL approach) for OA
* Ambulatory for a minimum of 10 meters with or without a mobility aid but without the assistance of another person
* Able to read, write and speak English
* Able to provide consent

Exclusion Criteria:

* Bilateral THA
* Underwent THA surgery for a diagnosis other than OA
* Any condition that will prevent participants from completing the study such as having a significant neurological, cardiovascular, musculoskeletal condition as denoted by their physician.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People receiving elective unilateral total hip arthroplasty for osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
The Balance Evaluation Systems Test (BESTest) | Pre-THA, and at 2, 6, and 12 weeks post-THA
  The BESTest is a comprehensive performance-based postural stability assessment tool. The BESTest consists of 36 items that assess each underlying component of the balance systems framework (i.e., static stability, motor systems, functional stability limits, verticality, reactive postural control, anticipatory postural control, dynamic stability, sensory integration, and cognitive influences). Each item is scored from 0 (severe balance impairment) to 3 (no balance impairment). The maximum total score is 108 points with higher scores representing better postural stability.
The Activities-specific Balance Confidence (ABC) scale | Pre-THA, and at 2, 6, and 12 weeks post-THA
  The 16-item ABC scale assesses the level of confidence a person has in performing a set of daily activities without losing their balance or feeling unsteady. The ABC scale evaluates balance confidence. Each item is rated on scale of 0% (no confidence) to 100% (complete confidence). The final score is the average of all 16-items. ABC scores can be categorized as follows: less than 50 is a low balance confidence, between 50 and 80 is a moderate balance confidence, and over 80 is a high balance confidence.

SECONDARY OUTCOMES:
The University of California, Los Angeles (UCLA) activity scale | Pre-THA, and at 2, 6, and 12 weeks post-THA
  The UCLA activity scale measures physical activity on a scale from 1 ("no physical activity, dependent on others") to 10 ("regular participation in impact sports"). It has been identified as the most suitable scale for assessing physical activity levels in people undergoing total joint arthroplasty.
The EuroQol-Five Dimensions-Five Levels (EQ-5D-5L) | Pre-THA, and at 2, 6, and 12 weeks post-THA
  The EQ-5D-5L is a generic preference-based measure that evaluates five dimensions of health-related quality of life: mobility, self-care, usual activities, pain/discomfort (PD), and anxiety/depression (AD). Each dimension has five response levels representing no, slight, moderate, severe, and extreme problems. In addition to the five dimensions, the EQ-5D-5L includes the EuroQol-visual analogue scales (EQ VAS), which allow individuals to rate their health status on a scale ranging from 0 (worst imaginable health) to 100 (best imaginable health). By using the Canadian EQ-5D-5L value set, health state utility values can be assigned to an EQ-described health state, ranging from -0.148 (representing 55,555) to 0.949 (representing 11,111). This is referred to as EQ-5D-5L utility.
The Harris Hip Score | Pre-THA, and at 2, 6, and 12 weeks post-THA
  The Harris Hip Score is an outcome measure completed by the surgeon and evaluates four domains related to the operated limb: pain, function, range of motion and absence of deformity. The score ranges from 0 (lowest outcome) to 100 (best outcome). Scoring can be interpreted as poor (<70), fair (70-79), good (80-89) or excellent (90-100).
The Western Ontario and McMaster Osteoarthritis Index (WOMAC) questionnaire | Pre-THA, and at 2, 6, and 12 weeks post-THA
  The WOMAC is a patient self-administered 24-item questionnaire divided into 3 subscales that assess pain, stiffness and joint function. For this study, a weighted and inverted conversion will be used for each domain with a maximum score of 100, where a higher score will indicate better overall health status.
Preoperative Fall Assessment: History of falls (previous 12 months), circumstances of falls, and injury (major or minor). | Pre-THA
  A history of fall questionnaire will be provided to participants to ascertain any falls that occurred in the previous 12 months before the THA surgery, circumstances of falls, and if any injuries occurred.
  A fall will be defined as an "unintentional coming to rest on the ground, floor or other lower level". Injuries will be categorized as major or minor. A major injury is defined as any fall that necessitates medical attention for the treatment of a fracture, while a minor injury is a bruise or laceration, where medical attention may or may not have been necessary.
Postoperative Fall Assessment: Prospective (daily) number of falls for 12 weeks post-THA, circumstances of falls, and injury (major or minor). | 2, 6, and 12 weeks post-THA
  Participants will be provided with a journal to record any falls (daily), circumstances of falls and information on any injuries. A face-to-face meeting will be conducted during their postoperative appointments to rectify any missing information. A fall will be defined as an "unintentional coming to rest on the ground, floor or other lower level". Injuries will be categorized as major or minor. A major injury is defined as any fall that necessitates medical attention for the treatment of a fracture, while a minor injury is a bruise or laceration, where medical attention may or may not have been necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Brent Lanting, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre- University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No